CLINICAL TRIAL: NCT02535078
Title: A Phase Ib/II Open-label, Multi-center Study of the Safety and Efficacy of IMCgp100 in Combination With Durvalumab (MEDI4736) or Tremelimumab or the Combination of Durvalumab and Tremelimumab Compared to IMCgp100 Alone in Patients With Advanced Melanoma
Brief Title: Phase 1b/2 Study of the Combination of IMCgp100 With Durvalumab and/or Tremelimumab in Advanced Cutaneous Melanoma
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Immunocore Ltd (Industry)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IMCgp100-201
Record Dates: First submitted 2015-08-26; First posted 2015-08-28 (Estimated); Last update posted 2024-07-24 (Actual); Status verified 2024-07

CONDITIONS: Malignant Melanoma
Keywords: IMCgp100; gp100; metastatic cutaneous melanoma; checkpoint inhibitor; PD-1; PD-L1; CTLA-4; durvalumab; tremelimumab; Tebentafusp; Bispecific T cell receptor fusion protein; ImmTAC; Immune mobilizing monoclonal T cell receptor against cancer; Immunotherapy; mucosal melanoma; acral melanoma; tebentafusp (IMCgp100); Kimmtrak
MeSH Terms: conditions — Melanoma; Diabetes Mellitus, Insulin-Dependent, 12 | interventions — tebentafusp

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Phase 2: Tebentafusp SC Monotherapy (Experimental): Tebentafusp (IMCgp100) (single agent) subcutaneous (SC) injection
  Interventions: Drug: Tebentafusp (IMCgp100)

INTERVENTIONS:
Drug: Tebentafusp (IMCgp100) — soluble gp100-specific T cell receptor with anti-CD3 scFV

SUMMARY:
This study was a mixed phase Ib/II, multi-center, open-label study of tebentafusp (IMCgp100) as a single agent, and in combination with durvalumab and/or tremelimumab, in metastatic cutaneous melanoma. The purpose of this study is to characterize the safety, tolerability, pharmacokinetics (PK), pharmacodynamics, and to evaluate the anti-tumor activity of tebentafusp (IMCgp100) in combination with durvalumab (MEDI4736, programmed death-ligand 1 [PD-L1] inhibitor), tremelimumab (CLTA-4 inhibitor), and the combination of durvalumab with tremelimumab compared to single-agent tebentafusp (IMCgp100) alone administered as an intravenous or subcutaneous. The study will enroll patients who have metastatic melanoma that is refractory to treatment with an anti-PD-1 inhibitor in the metastatic setting. This study will also evaluate the safety, tolerability, and anti-tumor activity of tebentafusp (IMCgp100) monotherapy in patients with advanced non-uveal melanoma who progressed on prior PD-1 inhibitors approved for the treatment of advanced melanoma; patients with BRAF mutations must be refractory to approved BRAF-based therapy.

DETAILED DESCRIPTION:
As of Amendment 9, a potential phase 2 portion of the study was to be opened after identification of the recommended phase 2 dose (RP2D) for Arm 5 (tebentafusp sc monotherapy). However, the phase 2 portion of the study was never initiated.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. Written informed consent must be obtained from all patients prior to any study procedures
3. Patients with advanced non-uveal melanoma defined as unresectable stage III or metastatic stage IV disease. Patients with acral or mucosal melanoma are acceptable. Patients with melanoma of unknown primary are acceptable for Phase 1b escalation cohorts (Arms 1 to 5) but are excluded in Phase 2. NOTE: Patients with the diagnosis of UM are excluded from all cohorts
4. Phase 1b (Arm 4 and Arm 5) and Phase 2: Patients with disease progression following initiation of treatment with an approved PD-(L)1 inhibitor. Patients with BRAF mutations should be refractory to approved BRAF-inhibitor if clinically feasible. CTLA 4 inhibition therapy is acceptable as a prior line of therapy or in combination with anti-PD-(L)1 therapy. For Phase 2, no prior chemotherapy in the advanced setting is permitted
5. Phase 1b Arms 1-3: no restriction on prior therapy
6. HLA-A*02:01 positive by central assay or by an 510K approved assay run in CLIA-certified laboratory
7. Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1
8. Life expectancy of at least 3 months
9. Phase 2 cohorts only: Patients must have measurable disease according to RECIST v1.1 criteria. Patients enrolled in Phase 1b cohorts may have either measurable or only non-measurable disease (ie, non-target lesion only)
10. Phase 1b (Arm 4) and Phase 2 cohorts only: Patients must have a site of disease amenable to biopsy (ie, must not also be a target lesion OR if a target lesion must be > 2cm), and be a candidate for tumor biopsy according to the treating institution's guidelines. NOTE: Phase 1b Arms 1-3 and 5 patients are not required to have disease accessible to biopsy
11. For Arms 1-3 only (ie, applies only to patients assigned to receive tebentafusp in combination with checkpoint inhibitor[s]): Those receiving prior immunotherapy must meet all the following conditions:

    1. Must not have experienced an immune-related adverse event (irAE) where the irAE was the reason for permanent discontinuation of prior immunotherapy in the most recent prior treatment regimen
    2. All irAEs while receiving prior immunotherapy must have resolved to ≤ Grade 1 or baseline prior to screening for this study. Must not have experienced a ≥ Grade 3 immune-related AE within the past 16 weeks or any Grade 4 life-threatening irAE (regardless of duration) or neurologic or ocular AE of any grade while receiving prior immunotherapy. (NOTE: Patients with endocrine AE of any grade are permitted to enroll if they are stably maintained on appropriate replacement therapy, but must have no history of adrenal crisis and be asymptomatic)
    3. Patients currently receiving chronic corticosteroid treatment (longer than 8 weeks duration) for management of pre-existing AEs, or patients with a history of chronic corticosteroid treatment longer than 8 weeks duration for AEs within 6 months of screening are excluded

Exclusion Criteria:

1. Presence of untreated or symptomatic central nervous system (CNS) metastases, leptomeningeal disease, or cord compression.
2. History of severe hypersensitivity reactions to study medications
3. History of treatment-related interstitial lung disease/pneumonitis
4. Impaired baseline organ function as evaluated by out-of-range laboratory values.
5. Clinically significant cardiac disease or impaired cardiac function
6. Active autoimmune disease or a documented history of autoimmune disease
7. Recent (< 12 months of planned first dose of study treatment) active diverticulitis (Phase 1b combination arms)
8. Active infection requiring systemic antibiotic therapy. NOTE: Patients requiring systemic antibiotics for infection must have completed therapy before planned first dose of study treatment
9. Known history of human immunodeficiency virus (HIV) infection. Testing for HIV status is not necessary unless clinically indicated or if required by local regulation
10. Active hepatitis B virus (HBV) or hepatitis C virus (HCV) infection, currently requiring medical intervention, per institutional protocol. Testing for HBV or HCV status is not necessary unless clinically indicated or the patient has a history of HBV or HCV infection requiring treatment with currently an unknown status. History of treated hepatitis is not exclusionary
11. Malignant disease, other than that being treated in this study. Exceptions to this exclusion include the following: malignancies that were treated curatively and have not recurred within 2 years after completion of treatment; completely resected basal cell and squamous cell skin cancers; any malignancy considered to be indolent and that has never required therapy; and completely resected carcinoma in situ of any type
12. Any medical condition that would, in the investigator's judgment, prevent the patient's participation in the clinical study due to safety concerns, compliance with clinical study procedures or interpretation of study results
13. Systemic anti-cancer therapy within 2 weeks of the planned first dose of study treatment. For cytotoxic agents that have major delayed toxicity and any prior immunotherapy approach, 3 weeks is indicated as washout period
14. Presence of NCI CTCAE ≥ Grade 2 toxicity (except alopecia, peripheral neuropathy, and ototoxicity, which are excluded if ≥ NCI CTCAE Grade 3) due to prior cancer therapy
15. Systemic treatment with steroids or any other immunosuppressive drug use within 4 weeks of the planned first dose of study treatment, with the following exceptions:

    1. Treatment for well-controlled and asymptomatic adrenal insufficiency is permitted, but replacement dosing is limited to prednisone ≤ 12 mg daily or the equivalent.
    2. Local steroid therapies (eg, optic, ophthalmic, intra-articular, or inhaled medications) are acceptable
    3. Premedication for allergy to contrast reagent or premedication regimen instituted per protocol
    4. Steroids for management of CNS metastases > 2 weeks prior to the planned first dose of study treatment
16. Use of any live vaccines against infectious diseases within 4 weeks of initiation of study treatment
17. Major surgery as defined by the investigator within 2 weeks of the first dose of study treatment.
18. Radiotherapy within 2 weeks of the first dose of study treatment, with the exception of palliative radiotherapy to a limited field, such as for the treatment of bone pain or a focally painful tumor mass
19. Use of hematopoietic colony-stimulating growth factors (eg, G-CSF, GMCSF, MCSF) ≤ 2 weeks prior start or study treatment. NOTE: Patients must have completed therapy with hematopoietic colony-stimulating factors at least 2 weeks before the first dose of study treatment is given. An erythroid stimulating agent is allowed as long as it was initiated at least 2 weeks prior to the first dose of study treatment and the patient is not red blood cell transfusion dependent
20. Pregnant or breast-feeding women
21. Women of child-bearing potential who are sexually active with a non-sterilized male partner, unless they are using highly effective contraception during study treatment, and must agree to continue using such precautions for 1 week after the final dose of investigational product; cessation of birth control after this point should be discussed with a responsible physician.
22. Male patients must be surgically sterile or use double barrier contraception method and are not allowed to donate sperm from enrollment through treatment and for 3 months following administration of the last dose of study drug
23. Patients who are relatives or dependents of the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2023-06-19 (Actual); Study Completion 2023-09-06 (Actual)

PRIMARY OUTCOMES:
Phase 2: Objective Response Rate (ORR) | Up to ~2 years

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - The Angeles Clinic and Research Institute, Los Angeles, California
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania

REFERENCES:
- [Derived] Hamid O, Hassel JC, Shoushtari AN, Meier F, Bauer TM, Salama AKS, Kirkwood JM, Ascierto PA, Lorigan PC, Mauch C, Orloff M, Evans TRJ, Holland C, Edukulla R, Abedin SE, Middleton MR. Tebentafusp in combination with durvalumab and/or tremelimumab in patients with metastatic cutaneous melanoma: a phase 1 study. J Immunother Cancer. 2023 Jun;11(6):e006747. doi: 10.1136/jitc-2023-006747. PMID 37286303